CLINICAL TRIAL: NCT00849849
Title: Comprehensive Postpartum Screening Strategies for Women With Prior Gestational Diabetes (COPSS - GDM): Now is the Time for a Paradigm Shift in Clinical Practice
Brief Title: Comprehensive Postpartum Screening Strategies for Women With Gestational Diabetes Mellitus (GDM)
Acronym: COPSS-GDM
Status: Completed | Type: Observational
Sponsor: Woman's (Other)
Responsible Party: Principal Investigator, Karen Elkind-Hirsch, Scientific Director of Research, Woman's
Other Study IDs: RO-08-11
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: postgestational diabetes; diabetes mellitus; OGTT; insulin sensitivity; insulin secretion
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for diabetes testing
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Postpartum GDM OGTT: 200 women with prior GDM in their index pregnancies will undergo postpartum screening assessment. This program will follow these women who are at a high risk of developing DM2 after delivery for 1 year.

SUMMARY:
Previous gestational diabetes (GDM) predisposes affected women to diabetes. Pregnancy, in essence, serves as a metabolic stress test and uncovers underlying insulin resistance and ß-cell dysfunction. Cumulative incidence rates of type 2 diabetes (DM2) among women with a history of GDM vary widely depending on the length of follow up and the underlying risk of diabetes in the population. Like DM2, the incidence of postpartum diabetes appears to be increasing The cumulative incidence of DM2 varied from 2.6 to > 70% in studies with postpartum follow-up ranging from 6 weeks to 28 years. Among women with a history of gestational diabetes, it is generally accepted that race, age, parity, family history of diabetes, pre-pregnancy weight, postpartum obesity, and weight gain are risk factors for developing DM2. Other suspected risk factors include smoking, physical inactivity, diet, and drugs that adversely affect glucose metabolism. Despite the high and increasing rate of DM2 in Louisiana, the medical community does not have reliable estimates of the number of woman living in southern Louisiana who develop diabetes subsequent to GDM. At Woman's Hospital, the investigators had 8246 deliveries in 2007; 7873 mothers (95% of deliveries) were either African American or Caucasian. Of this group of women, 665 were diagnosed with gestational diabetes mellitus. Thus, around 8.5% of the African American and Caucasian women delivering babies at Woman's Hospital in 2007 had a glucose abnormality. The incidence of diabetes and impaired glucose metabolism in the immediate postpartum period and within 12 months after delivery in this population is unknown. There are no long-term studies performed in Louisiana that have compared the benefits of different screening strategies or evaluated an optimum testing frequency after GDM to reduce the rate of DM2 and cardiovascular disease (CVD) in these high-risk women. The investigators plan to use this study as an outreach effort to provide screening for previous gestational diabetic mothers without adequate medical coverage following delivery.

DETAILED DESCRIPTION:
Women with previous gestational diabetes constitute an ideal group for the development, testing, and implementation of clinical strategies for primary diabetes prevention. One-third to one-half of women with a history of GDM will develop type 2 (DM2) within 3-5 years and 70% will develop DM2 if followed >10 years. Studies have shown that measuring only the fasting glucose level postpartum is not sufficiently sensitive to identify all women who have impaired glucose tolerance (IGT) or DM2. Data presented at the Fifth International Workshop-Conference on GDM indicated that, postpartum, only 34% of the women with IGT or DM2 had impaired fasting glucose and that 44% of those with DM2 had fasting levels below 100 mg/dl (<5.5 mmol/l). The recommended process to detect permanent diabetes in women who have had GDM and who might become pregnant again is a 75-g 2-h oral glucose tolerance test (OGTT) 6-12 weeks post partum and every year thereafter. Postpartum management of women with GDM is critical because of their markedly increased risk of DM2 and its comorbidities in the future Follow-up studies of women with GDM are necessary to establish the most efficient and most-effective approach to postpartum screening for type 2 diabetes. This study will examine the diagnostic effectiveness of OGTT-derived glucose tolerance, insulin secretion and insulin sensitivity indices compared with indices derived from fasting values of glucose and insulin in subjects with GDM performed post-partum. We will establish whether post-partum fasting and/or glucose-stimulated indices of insulin sensitivity and secretion most accurately estimate the degree of insulin resistance relative to ß-cell function in all race/ethnicity groups of women after delivery of a pregnancy complicated by gestational diabetes and predict their risk for development of diabetes and CVD. .Primary Objective1) We will identify, recruit and test 100 individuals with prior GDM in order to:§ Determine the best way to assess glucose tolerance disorders' prevalence after pregnancy complicated by GDM in southern Louisiana.§ Determine the most effective screening strategy to identify those women with prior GDM who develop or are at high risk for developing DM2 and comorbidities postpartum.A 2 hr, 75-gram OGTT with measurements of insulin and glucose will be performed at their 6-12 week and 1-year post-delivery check-up; this will be compared with the results of their single fasting glucose and insulin value.Secondary Objectives1) We will measure cardiometabolic markers (lipids, blood pressure) in the COPS-GDM study in order to:§ Identify the frequency and value of CVD risk markers in women with glucose abnormalities persisting after pregnancies with GDMGlucometabolic perturbations carry a particularly high risk for metabolic syndrome in women with prior GDM. Woman with prior GDM shown to have higher blood pressure and an altered lipid profile with increased LDL cholesterol and triglyceride levels and decreased HDL cholesterol levels that correlate with cardiovascular disease (CVD) risk factors2) We will measure anthropometric measures (body weight, BMI, abdominal girth) and liver aminotransferase levels (ALT, AST) in order to:§ Determine if there is a higher prevalence of postpartum glucose abnormalities in women with prior GDM predicted by BMI category and/or abdominal adiposity § Determine if elevated abnormal aminotransferase activity is more prominent in prior GDM women and the relationship to subsequent diabetes Former gestational diabetic mothers when compared with women with no history of GDM are found to have higher body mass index (BMI) and visceral adiposity. The distribution of postpartum glucose abnormalities by BMI category was found to be more common with increased BMI.3) We will investigate the impact of breastfeeding in women with a prior GDM on glucose tolerance and CVD risk factors to:§ Determine if lactation has immediate and long-term favorable effects in this patient population postpartum.Breast-feeding has been associated with significantly lower triglyceride level, higher HDL cholesterol, lower total cholesterol/HDL ratio, lower mean fasting glucose, and lower prevalence of any postpartum abnormality of glucose tolerance, including diabetes. Breastfeeding has also been reported to lower the rate of overt diabetes developing later in life in women with a history of gestational diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum Women (6-12 weeks)who experienced GDM during index pregnancy 18 years to 42 years of age
* English-speaking
* Written consent for participation in the study

Exclusion Criteria (Medical):

* Cholestasis during the past pregnancy
* Serum AST and/or ALT level exceeding more than twice normal laboratory values
* History or clinical manifestation of cardiovascular disease
* History or clinical manifestation of diabetes or use of anti-diabetic drugs before pregnancy
* History or clinical manifestation of any other significant metabolic, hematologic, pulmonary, cardiovascular, gastrointestinal, neurologic, immune, hepatic, renal, urologic disorders, or cancer
* Regular use of medications for weight control, psychosis and hormonal birth control
* Current use of medication to treat diabetes

Exclusion Criteria (Psychiatric and Behavioral):

* History or clinical manifestation of any eating disorder
* Individuals who smoke
* History of drug or alcohol abuse (up to 14 drinks a week are allowed) within the past two years

Other Exclusion Criteria:

* Pregnancy or pregnancy planned during the coming year
* Not willing or unable to adhere to the clinical evaluation schedule over the twelve -month study period

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Postpartum women with GDM (before 12 weeks postpartum)
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Determine best way to assess glucose disorder prevalence in women with prior GDM | 3 years
  A 2 hr, 75-gram OGTT with measurements of insulin and glucose will be performed at their 6-12 week and 1-year post-delivery check-up; this will be compared with the results of their single fasting glucose and insulin value.

SECONDARY OUTCOMES:
Investigate if cardiometabolic markers-lipid profile and blood pressure anthropometric markers such as BMI [BMI, absolute body weight]; visceral adiposity as assessed by abdominal girth are associated with an increased diabetes risk | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Elkind-Hirsch, MSc,PhD, Principal Investigator — Woman's Health Research Institute
Locations (1):
- Woman's Hospital Research Institute, Baton Rouge, Louisiana, United States